CLINICAL TRIAL: NCT06414278
Title: Early Identification of Cognitive Side-Effects of Immunotherapy
Brief Title: Evaluation of Early Identification of Cognitive Side Effects of Immunotherapy
Status: Recruiting | Type: Observational
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2022LS089; NCI-2023-09048 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2022LS089 (Other: University of Minnesota/Masonic Cancer Center); P30CA077598 (NIH)
Record Dates: First submitted 2024-05-08; First posted 2024-05-16 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients complete SALSA assessment and ICE assessments on study. Patients also have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This clinical trial evaluates the use of a tool kit, Stress, Affect, Language and Speech Analysis (SALSA), for early identification of cognitive side effects of immunotherapy compared to the standard of care assessment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate the use of a toolkit for automated administration and scoring of cognitive tests (Stress, Language and Speech Analysis, or SALSA) in adult cancer patients who are treated with commercial chimeric antigen receptor T cell therapy (CAR-T) products at University of Minnesota and are at risk of developing immune effector cell-associated neurotoxicity syndrome (ICANS).

OUTLINE: This is an observational study.

Patients complete SALSA assessment and ICE assessments on study. Patients also have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* * ≥ 18 years of age at initiation of therapy

  * Planning to undergo inpatient CAR-T therapy for primary malignancy
  * Fluent in English (written or spoken)

Exclusion Criteria:

* * Subjects with speech or hearing impediment that would make them unable to be assessed with SALSA

  * Subjects with diagnosed cognitive impairment prior to CAR-T therapy
  * Unwilling or unable to sign voluntary written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients planning to undergo CAR-T therapy for primary malignancy recruited through the University of Minnesota.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2027-07-21 (Estimated); Study Completion 2028-02-21 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients completing at least 80 percent of planned SALSA administrations during post CAR-T hospitalization | 18 months
  Descriptive statistics will be used to summarize the feasibility of SALSA in CAR-T patients. The overall completion rate of will be calculated for each patient, as well as the pattern of completions.

CONTACTS AND LOCATIONS:
Overall Officials: Veronika Bachanova, Principal Investigator — University of Minnesota Masonic Cancer Center
Locations (1):
- University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota, United States